CLINICAL TRIAL: NCT06514859
Title: Outcomes of Laparoscopic Versus Open Repair of Inguinal Hernia
Brief Title: Repair of Inguinal Hernia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abdelaziz Mohamed Abdelaziz, Resident at General, Oncology, Laparoscopic Surgery Department , Faculty of Medicine, Sohag University, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-06-07MS
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-06

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic repair of inguinal hernia (Active Comparator)
  Interventions: Procedure: Laparoscopic repair of inguinal hernia
- Open repair of inguinal hernia (Active Comparator)
  Interventions: Procedure: Open repair of inguinal hernia

INTERVENTIONS:
Procedure: Laparoscopic repair of inguinal hernia — Laparoscopic repair of inguinal hernia
  Arms: Laparoscopic repair of inguinal hernia
Procedure: Open repair of inguinal hernia — Repair of inguinal hernia by open technique-mesh hernioplasty -
  Arms: Open repair of inguinal hernia

SUMMARY:
The aim of this study is to compare the outcomes of open versus laparoscopic approaches for inguinal hernia surgery and provide evidence-based guidance to the selection of the most appropriate operative technique.

ELIGIBILITY:
Inclusion Criteria:

Male patient > 18 years of age

• Primary groin hernias requiring surgical intervention that are eligible for both open and laparoscopic repair.

Exclusion Criteria:

* Emergency procedures .

  * ASA score > 2.
  * Irreducible inguinoscrotal hernia .
  * Local or systemic infection .
  * Other abdominal hernias being operated at the same time or planned operated during Follow up.

Previous surgery which has impaired the sensation in the groin area .

* BMI > 40 kg/m2.
* Known disease which Impairs central or peripheral nerve function .
* Concurrent malignant Disease .
* Chronic pain which requires daily medication . • Mental disorder which requires daily medication .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence in management of inguinal hernia | 6 months after operation
  Rate of recurrence in both open and laparoscopic repair of inguinal hernia

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Bhandarkar DS, Shankar M, Udwadia TE. Laparoscopic surgery for inguinal hernia: Current status and controversies. J Minim Access Surg. 2006 Sep;2(3):178-86. doi: 10.4103/0972-9941.27735. PMID 21187993
- [Background] Aguirre DA, Casola G, Sirlin C. Abdominal wall hernias: MDCT findings. AJR Am J Roentgenol. 2004 Sep;183(3):681-90. doi: 10.2214/ajr.183.3.1830681. No abstract available. PMID 15333356
- [Background] McCormack K, Wake B, Perez J, Fraser C, Cook J, McIntosh E, Vale L, Grant A. Laparoscopic surgery for inguinal hernia repair: systematic review of effectiveness and economic evaluation. Health Technol Assess. 2005 Apr;9(14):1-203, iii-iv. doi: 10.3310/hta9140. PMID 15842951